CLINICAL TRIAL: NCT03757130
Title: A Phase 1b, Randomized, Double-blind, Placebo-controlled, Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AMG 598 in Subjects With Obesity
Brief Title: Multiple Ascending Dose Study of AMG 598 in Adults With Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: 20170139
Record Dates: First submitted 2018-11-27; First posted 2018-11-28 (Actual); Results first posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2022-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Placebo (Placebo Comparator): Participants received placebo subcutaneous injection once every 4 weeks (Q4W) for a total of 3 doses.
  Interventions: Drug: Placebo
- Placebo + Liraglutide (Active Comparator): Participants received placebo subcutaneous injection once every 4 weeks for a total of 3 doses in addition to liraglutide administered by subcutaneous injection once a day for 12 weeks. The starting dose of liraglutide was 0.6 mg/day, increasing in increments of 0.6 mg/day every 7 days to reach the full dosage of 3 mg/day by week 5.
  Interventions: Drug: Placebo; Drug: Liraglutide
- AMG 598 70 mg (Experimental): Participants received 70 mg AMG 598 by subcutaneous injection once every 4 weeks (Q4W) for a total of 3 doses.
  Interventions: Drug: AMG 598
- AMG 598 70 mg + Liraglutide (Experimental): Participants received 70 mg AMG 598 by subcutaneous injection once every 4 weeks for a total of 3 doses in addition liraglutide administered by subcutaneous injection once a day for 12 weeks. The starting dose of liraglutide was 0.6 mg/day, increasing in increments of 0.6 mg/day every 7 days to reach the full dosage of 3 mg/day by week 5.
  Interventions: Drug: AMG 598; Drug: Liraglutide
- AMG 598 210 mg (Experimental): Participants received 210 mg AMG 598 by subcutaneous injection once every 4 weeks for a total of 3 doses.
  Interventions: Drug: AMG 598
- AMG 598 210 mg + Liraglutide (Experimental): Participants received 210 mg AMG 598 by subcutaneous injection once every 4 weeks for a total of 3 doses in addition to liraglutide administered by subcutaneous injection once a day for 12 weeks. The starting dose of liraglutide was 0.6 mg/day, increasing in increments of 0.6 mg/day every 7 days to reach the full dosage of 3 mg/day by week 5.
  Interventions: Drug: AMG 598; Drug: Liraglutide
- AMG 598 420 mg (Experimental): Participants received 420 mg AMG 598 by subcutaneous injection once every 4 weeks for a total of 3 doses.
  Interventions: Drug: AMG 598
- AMG 598 420 mg + Liraglutide (Experimental): Participants received 420 mg AMG 598 by subcutaneous injection once every 4 weeks for a total of 3 doses in addition to liraglutide administered by subcutaneous injection once a day for 12 weeks. The starting dose of liraglutide was 0.6 mg/day, increasing in increments of 0.6 mg/day every 7 days to reach the full dosage of 3 mg/day by week 5.
  Interventions: Drug: AMG 598; Drug: Liraglutide

INTERVENTIONS:
Drug: AMG 598 — AMG 598 administered by subcutaneous injection
  Arms: AMG 598 210 mg; AMG 598 210 mg + Liraglutide; AMG 598 420 mg; AMG 598 420 mg + Liraglutide; AMG 598 70 mg; AMG 598 70 mg + Liraglutide
Drug: Placebo — Placebo matching to AMG 598 administered by subcutaneous injection
  Arms: Placebo; Placebo + Liraglutide
Drug: Liraglutide — Liraglutide administered by subcutaneous injection. The starting dose is 0.6 mg/day, and increased by 0.6 mg/day dose increment every 7 days, up to the full dosage of 3.0 mg/day by week 5.
  Other Names: Saxenda®
  Arms: AMG 598 210 mg + Liraglutide; AMG 598 420 mg + Liraglutide; AMG 598 70 mg + Liraglutide; Placebo + Liraglutide

SUMMARY:
The main objective of this study is to assess the safety and tolerability of multiple doses of AMG 598 administered alone or in combination with liraglutide in adults with obesity.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with ages between 18 and 65 years old, inclusive, at time of signing consent
* Body mass index (BMI) between greater than or equal to 30.0 kg/m^2 and less than or equal to 40.0 kg/m^2 at screening
* Except for obesity, otherwise healthy or medically stable per protocol
* Have a stable body weight defined as less than 5 kg self-reported change during the previous 8 weeks prior to screening
* Other Inclusion criteria may apply
* Stable on liraglutide, depending on cohort

Exclusion Criteria:

* History or clinical evidence of diabetes
* Inadequate organ function at screening
* Currently receiving treatment in another investigational device or drug study
* Women who are pregnant/lactating/breastfeeding or who plan to become pregnant/breastfeed while on study through 5 months after receiving the last dose of investigational product
* History or evidence of a clinically significant disorder, condition or disease that would pose a risk to subject safety or interfere with the study evaluation, procedures or completion
* A family or personal history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2; a personal history of non-familial medullary thyroid carcinoma; confirmed chronic pancreatitis or idiopathic acute pancreatitis, or gallbladder disease (ie, cholelithiasis or cholecystitis) not treated with cholecystectomy, for cohorts receiving liraglutide
* History of major depressive disorder
* Other Exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (4):
- United States (4):
  - William D Summers MD LLC, Birmingham, Alabama
  - Orange County Research Center, Tustin, California
  - QPS Miami Research Associates, South Miami, Florida
  - Dallas Diabetes and Endocrine Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 2 centers in the United States.
Pre-assignment Details: Eligible participants were randomized to one of six treatment cohorts. Within each cohort participants were randomly assigned in a 3:1 ratio to receive either AMG 598 or placebo.
Period: Overall Study
Arm/Group | Placebo | Placebo + Liraglutide | AMG 598 70 mg | AMG 598 70 mg + Liraglutide | AMG 598 210 mg | AMG 598 210 mg + Liraglutide | AMG 598 420 mg | AMG 598 420 mg + Liraglutide
Started | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 7 | 6 | 6 | 5 | 5
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Placebo + Liraglutide | AMG 598 70 mg | AMG 598 70 mg + Liraglutide | AMG 598 210 mg | AMG 598 210 mg + Liraglutide | AMG 598 420 mg | AMG 598 420 mg + Liraglutide | Total
Number analyzed (Participants) | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (11.0) | 41.8 (7.6) | 41.7 (11.3) | 46.1 (14.2) | 50.3 (7.8) | 51.5 (8.5) | 44.5 (10.9) | 49.2 (11.7) | 46.5 (10.6)
Age, Customized [Count of Participants; unit: Participants]
  < 40 years | 1 | 2 | 3 | 3 | 1 | 1 | 2 | 1 | 14
  ≥ 40 years | 5 | 4 | 3 | 5 | 5 | 5 | 4 | 5 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 1 | 4 | 3 | 3 | 1 | 1 | 15
  Male | 4 | 6 | 5 | 4 | 3 | 3 | 5 | 5 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 4 | 8 | 6 | 6 | 3 | 5 | 41
  Not Hispanic or Latino | 2 | 1 | 2 | 0 | 0 | 0 | 3 | 1 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 3 | 1 | 1 | 2 | 1 | 1 | 10
  White | 5 | 6 | 3 | 7 | 5 | 3 | 5 | 5 | 39
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 34.22 (2.61) | 33.20 (2.10) | 34.62 (2.92) | 35.46 (2.19) | 34.43 (3.37) | 34.42 (3.24) | 32.77 (3.04) | 36.00 (4.04) | 34.43 (2.92)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: The investigator assessed the severity of each adverse event reported during the study. The assessment was based on the Amgen Standard Grading Scale:
  Mild: Aware of sign or symptom, but easily tolerated. Moderate: Discomfort enough to cause interference with usual activity. Severe: Incapacitating with inability to work or do usual activity.
  A Serious adverse event is defined as any untoward medical occurrence that, met at least 1 of the following serious criteria
  * Death;
  * Was life-threatening;
  * Required in-patient hospitalization or prolongation of existing hospitalization;
  * Resulted in persistent or significant disability/incapacity;
  * Was a congenital anomaly/birth defect;
  * Other medically important serious event.
  The investigator also assessed whether each adverse event was related to study drug administration based on clinical judgement.
Time Frame: 207 days
Population: All participants who received at least 1 dose of study drug (AMG 598 or placebo) on day 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Placebo + Liraglutide | AMG 598 70 mg | AMG 598 70 mg + Liraglutide | AMG 598 210 mg | AMG 598 210 mg + Liraglutide | AMG 598 420 mg | AMG 598 420 mg + Liraglutide
Number analyzed (Participants) | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6
Participants
  All treatment-emergent adverse events (TEAEs) | 1 | 6 | 4 | 7 | 5 | 6 | 0 | 4
  Mild TEAEs | 1 | 6 | 4 | 7 | 5 | 6 | 0 | 4
  Moderate TEAEs | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1
  Severe TEAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Serious TEAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  TEAE leading to discontinuation of AMG 598 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  TEAE leading to discontinuation of liraglutide | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
  Life-threatening TEAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fatal TEAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Maximum Observed Concentration (Cmax) of AMG 598 After Subcutaneous Injection on Day 1 and Day 57
Description: Serum concentrations of AMG 598 were determined using a validated electrochemiluminescence-based method. The lower limit of quantitation was 50.0 ng/mL.
Time Frame: Day 1, predose, and days 6, 8, 15, 22, and 29; Day 57 predose and days 62, 64, 71, 85, 99, 113, 127, 169, and 207
Population: The pharmacokinetic (PK) analysis set included all participants for whom at least 1 PK parameter or endpoint could be adequately estimated. Participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | AMG 598 70 mg | AMG 598 70 mg + Liraglutide | AMG 598 210 mg | AMG 598 210 mg + Liraglutide | AMG 598 420 mg | AMG 598 420 mg + Liraglutide
Number analyzed (Participants) | 6 | 8 | 6 | 6 | 6 | 6
µg/mL
  Day 1 | 5.83 (1.67) | 7.49 (1.17) | 21.5 (5.43) | 18.0 (5.76) | 51.1 (9.70) | 36.9 (13.7)
  Day 57: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5
  Day 57 | 9.07 (1.91) | 12.0 (2.56) | 45.4 (12.5) | 34.8 (12.0) | 93.2 (18.2) | 72.4 (23.0)

3. Primary Outcome: Number of Participants With TEAEs Due to Laboratory, Electrocardiogram, and Vital Sign Findings
Description: TEAEs due to laboratory, electrocardiogram (ECG) and vital sign findings include any abnormal laboratory test results (hematology, clinical chemistry, or urinalysis) or electrocardiogram, or vital signs measurements, including those that worsened from baseline, that were considered clinically significant in the medical and scientific judgment of the investigator (ie, not related to progression of underlying disease).
Time Frame: 207 days
Population: All participants who received at least 1 dose of study drug (AMG 598 or placebo) on day 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Placebo + Liraglutide | AMG 598 70 mg | AMG 598 70 mg + Liraglutide | AMG 598 210 mg | AMG 598 210 mg + Liraglutide | AMG 598 420 mg | AMG 598 420 mg + Liraglutide
Number analyzed (Participants) | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6
Participants
  Blood creatine phosphokinase increased | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Electrocardiogram T wave abnormal | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hepatic enzyme increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Lipase increased | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 1
  Hypertension | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Time to Maximum Observed Concentration (Tmax) of AMG 598 After Subcutaneous Injection on Day 1 and Day 57
Description: as for outcome 2
Time Frame: Day 1, predose, and days 6, 8, 15, 22, and 29; Day 57 predose and days 62, 64, 71, 85, 99, 113, 127, 169, and 207
Population: The PK analysis set; participants with available data at each time point
Measure: Median (Full Range); unit: days
Arm/Group | AMG 598 70 mg | AMG 598 70 mg + Liraglutide | AMG 598 210 mg | AMG 598 210 mg + Liraglutide | AMG 598 420 mg | AMG 598 420 mg + Liraglutide
Number analyzed (Participants) | 6 | 8 | 6 | 6 | 6 | 6
days
  Day 1 | 7.1 [7.1 to 14] | 7.0 [5.0 to 21] | 7.1 [5.0 to 13] | 7.0 [4.9 to 14] | 6.9 [5.0 to 7.3] | 7.0 [6.9 to 14]
  Day 57: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5
  Day 57 | 7.0 [7.0 to 14] | 7.0 [7.0 to 7.0] | 6.1 [5.1 to 7.0] | 6.5 [5.0 to 8.0] | 5.3 [4.3 to 8.0] | 7.0 [7.0 to 11]

5. Secondary Outcome: Dose-normalized Cmax of AMG 598 After Subcutaneous Injection on Day 1 and Day 57
Description: as for outcome 2
Time Frame: Day 1, predose, and days 6, 8, 15, 22, and 29; Day 57 predose and days 62, 64, 71, 85, 99, 113, 127, 169, and 207
Population: The PK analysis set; participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: µg/mL/mg
Arm/Group | AMG 598 70 mg | AMG 598 70 mg + Liraglutide | AMG 598 210 mg | AMG 598 210 mg + Liraglutide | AMG 598 420 mg | AMG 598 420 mg + Liraglutide
Number analyzed (Participants) | 6 | 8 | 6 | 6 | 6 | 6
µg/mL/mg
  Day 1 | 0.0833 (0.0239) | 0.107 (0.0167) | 0.102 (0.0258) | 0.0856 (0.0274) | 0.122 (0.0231) | 0.0879 (0.0327)
  Day 57: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5
  Day 57 | 0.130 (0.0272) | 0.172 (0.0366) | 0.216 (0.0593) | 0.168 (0.0572) | 0.222 (0.0433) | 0.172 (0.05949)

6. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to 28 Days (AUC0-28) for AMG 598 After Subcutaneous Injection on Day 1 and Day 57
Description: as for outcome 2
Time Frame: Day 1, predose, and days 6, 8, 15, 22, and 29; Day 57 predose and days 62, 64, 71, and 85
Population: The PK analysis set; participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: days*µg/mL
Arm/Group | AMG 598 70 mg | AMG 598 70 mg + Liraglutide | AMG 598 210 mg | AMG 598 210 mg + Liraglutide | AMG 598 420 mg | AMG 598 420 mg + Liraglutide
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 6 | 6
days*µg/mL
  Day 1: number analyzed (Participants) | 4 | 6 | 5 | 5 | 6 | 5
  Day 1 | 139 (19.6) | 147 (21.8) | 495 (72.7) | 366 (101) | 1080 (225) | 763 (285)
  Day 57: number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 5
  Day 57 | 215 (45.3) | 276 (57.6) | 964 (203) | 749 (254) | 1990 (341) | 1610 (511)

7. Secondary Outcome: Dose-normalized AUC0-28 for AMG 598 After Subcutaneous Injection on Day 1 and Day 57
Description: as for outcome 2
Time Frame: Day 1, predose, and days 6, 8, 15, 22, and 29; Day 57 predose and days 62, 64, 71, and 85
Population: The PK analysis set; participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: days*µg/mL/mg
Arm/Group | AMG 598 70 mg | AMG 598 70 mg + Liraglutide | AMG 598 210 mg | AMG 598 210 mg + Liraglutide | AMG 598 420 mg | AMG 598 420 mg + Liraglutide
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 6 | 6
days*µg/mL/mg
  Day 1: number analyzed (Participants) | 4 | 6 | 5 | 5 | 6 | 5
  Day 1 | 1.98 (0.279) | 2.10 (0.311) | 2.36 (0.346) | 1.74 (0.480) | 2.57 (0.535) | 1.82 (0.680)
  Day 57: number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 5
  Day 57 | 3.07 (0.647) | 3.94 (0.823) | 4.59 (0.966) | 3.57 (1.21) | 4.75 (0.812) | 3.84 (1.22)

8. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to Time of Last Quantifiable Concentration (AUClast) of AMG 598 After Subcutaneous Injection on Day 57
Description: as for outcome 2
Time Frame: Day 57 predose and days 62, 64, 71, 85, 99, 113, 127, 169, and 207
Population: The PK analysis set; participants with available data for AUClast.
Measure: Mean (Standard Deviation); unit: days*µg/mL
Arm/Group | AMG 598 70 mg | AMG 598 70 mg + Liraglutide | AMG 598 210 mg | AMG 598 210 mg + Liraglutide | AMG 598 420 mg | AMG 598 420 mg + Liraglutide
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5
days*µg/mL | 458 (102) | 612 (129) | 2130 (334) | 1570 (462) | 4060 (1610) | 3060 (920)

9. Secondary Outcome: Accumulation Ratio (AR) for Cmax of AMG 598 After Subcutaneous Injection on Day 1 and Day 57
Description: Serum concentrations of AMG 598 were determined using a validated electrochemiluminescence-based method. The lower limit of quantitation was 50.0 ng/mL.
  Accumulation ratio for Cmax = Day 57 Cmax / Day 1 Cmax.
Time Frame: Day 1, predose, and days 6, 8, 15, 22, and 29; Day 57 predose and days 62, 64, 71, 85, 99, 113, 127, 169, and 207
Population: The PK analysis set; participants with available data at both time points.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | AMG 598 70 mg | AMG 598 70 mg + Liraglutide | AMG 598 210 mg | AMG 598 210 mg + Liraglutide | AMG 598 420 mg | AMG 598 420 mg + Liraglutide
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5
ratio | 1.62 (0.394) | 1.70 (0.237) | 2.12 (0.251) | 1.92 (0.207) | 1.83 (0.138) | 2.13 (0.418)

10. Secondary Outcome: Accumulation Ratio of AUC0-28 for AMG 598 After Subcutaneous Injection on Day 1 and Day 57
Description: Serum concentrations of AMG 598 were determined using a validated electrochemiluminescence-based method. The lower limit of quantitation was 50.0 ng/mL.
  The accumulation ratio for AUC0-28 = Day 57 AUC0-28 / Day 1 AUC0-28.
Time Frame: Day 1, predose, and days 6, 8, 15, 22, and 29; Day 57 predose and days 62, 64, 71, and 85
Population: The PK analysis set; participants with available data at both time points.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | AMG 598 70 mg | AMG 598 70 mg + Liraglutide | AMG 598 210 mg | AMG 598 210 mg + Liraglutide | AMG 598 420 mg | AMG 598 420 mg + Liraglutide
Number analyzed (Participants) | 4 | 5 | 5 | 5 | 5 | 4
ratio | 1.74 (0.480) | 1.84 (0.223) | 2.09 (0.254) | 1.86 (0.186) | 1.96 (0.177) | 2.17 (0.291)

11. Secondary Outcome: Terminal Half-life (T1/2,z) of AMG 598 After Subcutaneous Injection on Day 57
Description: as for outcome 2
Time Frame: Day 57 predose and days 62, 64, 71, 85, 99, 113, 127, 169, and 207
Population: The PK analysis set; participants with available data for T1/2,z
Measure: Mean (Standard Deviation); unit: days
Arm/Group | AMG 598 70 mg | AMG 598 70 mg + Liraglutide | AMG 598 210 mg | AMG 598 210 mg + Liraglutide | AMG 598 420 mg | AMG 598 420 mg + Liraglutide
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 5
days | 28.2 (3.04) | 31.5 (6.05) | 35.2 (5.86) | 29.1 (3.02) | 35.8 (3.21) | 29.8 (6.72)

ADVERSE EVENTS:
Time Frame: From first dose of AMG 598/placebo through the end of study; 207 days.
Groups:
- AMG 598 70 mg: Participants received 70 mg AMG 598 by subcutaneous injection once every 4 weeks for a total of 3 doses.
Arm/Group | Placebo | Placebo + Liraglutide | AMG 598 70 mg | AMG 598 70 mg + Liraglutide | AMG 598 210 mg | AMG 598 210 mg + Liraglutide | AMG 598 420 mg | AMG 598 420 mg + Liraglutide
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/8 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/8 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/6 | 6/6 | 4/6 | 7/8 | 5/6 | 6/6 | 0/6 | 4/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=6) | Placebo + Liraglutide (N=6) | AMG 598 70 mg (N=6) | AMG 598 70 mg + Liraglutide (N=8) | AMG 598 210 mg (N=6) | AMG 598 210 mg + Liraglutide (N=6) | AMG 598 420 mg (N=6) | AMG 598 420 mg + Liraglutide (N=6)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 4 | 1 | 2 | 1 | 2 | 0 | 3
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 2
Early satiety (General disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 1
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site haematoma (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site haemorrhage (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Furuncle (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 1 | 2 | 3 | 4 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram T wave abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 4 | 0 | 5 | 1 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2019-06-25): https://cdn.clinicaltrials.gov/large-docs/30/NCT03757130/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-22): https://cdn.clinicaltrials.gov/large-docs/30/NCT03757130/SAP_001.pdf